CLINICAL TRIAL: NCT03653468
Title: Similar Improvements in Cardiometabolic Risk Factors for Preventing the Metabolic Syndrome in Latinoamerican Amerindians After 12-weeks of Concurrent Training
Brief Title: Exercise for Preventing the Metabolic Syndrome in Latinoamerican Amerindians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad del Rosario (Other); Universidad Pública de Navarra (Other); Healthcare Center Tomas Rojas (Other); Universidad de Los Lagos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 28082018
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Cardiovascular Risk Factor; Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Behavioral
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No-exercise
- Endurance training plus resistant training (Experimental): Concurrent training
  Interventions: Behavioral: Concurrent training (CT)

INTERVENTIONS:
Behavioral: Concurrent training (CT) — The core part of each session included resistance training (RT) followed by aerobic training exercises (for 50 and 30 minutes, respectively) and was preceded and followed by a 5-minute warm-up and cool-down with callisthenic movements.
  Arms: Endurance training plus resistant training

SUMMARY:
Despite exercise training decrease blood fasting glicaemy in 'average' terms, there is a wide inter-individual variability after exercise training explored mainly in adults but not in adults with prediabetes comorbidities. Thus, is yet unknown the effects and influence of the concurrent training (CT) eliciting responders (R) and non-responders (NR) cases (i.e., percentage of subjects who experienced a non-change/worsened response after training in some metabolic outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Interested in improving health and fitness

Exclusion Criteria:

* Cardiovascular contraindications to exercise
* History of stroke, asthma or chronic obstructive pulmonary disease, muscle-skeletal disorders
* Smoking
* A compliance rate to the exercise program ≥ 70% was required for the participants in the intervention group to be included in the statistical analyses.

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in fasting glucose
Total cholesterol | Baseline and 20-weeks immediately after the interventions ends
  Change from baseline in Total cholesterol
Blood pressure | Baseline and 20-weeks immediately after the interventions ends
  Change from baseline in Blood pressure

SECONDARY OUTCOMES:
Body mass | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in body mass
Waist circumference | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in waist circumference
Fat mass | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in fat mass
Lean mass | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in lean mass
Heart rate at rest | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in heart rate at rest
Six minutes walking test | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in six minutes walking test

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Alvarez, PhD, Principal Investigator — Universidad de Los Lagos
Locations (1):
- Cristian Alvarez, Los Lagos, Osorno, Chile

IPD SHARING:
Plan to Share IPD: No
Statistical Analysis Plan